CLINICAL TRIAL: NCT03651167
Title: Skin Tone Preferences and Their Influence on Skin Care Behaviors
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Roopal Kundu, Principal Investigator, Northwestern University
Other Study IDs: RVK05222018
Record Dates: First submitted 2018-08-27; First posted 2018-08-29 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Dermatology/Skin - Other
Keywords: skin care; skin tone; tanning; skin tone preference
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey — Participants will complete a survey online

SUMMARY:
The purpose of this study is to classify participants by actual skin tone and skin tone preference and identify whether an association exists between these skin tone preferences and knowledge of skin care recommendations, attitudes towards healthy skin care, or skin care behaviors.

DETAILED DESCRIPTION:
This study seeks to examine if there is a difference between ideal and actual skin tone among minority populations. In addition, we hope to assess whether various demographic factors as well as disparity between ideal and actual skin tone effect skin protective behaviors (i.e. sun screen use, dermatologist appointments, skin self-exams) or skin destructive behaviors (i.e. outdoor tanning, tanning salon use, use of skin lightening products) in minority populations.

ELIGIBILITY:
Inclusion Criteria:

* Subjects age 18 years old or older
* Self-identified members of a minority (African, Asian, Hispanic/Latino, American Indian, Alaskan native, etc.) population
* Subjects who are capable of completing an online, English survey

Exclusion Criteria:

* Subjects age 17 years old or younger
* Subjects not self-identified members of a minority (African, Asian, Hispanic/Latino, American Indian, Alaskan native, etc.) population
* Subjects who are incapable of completing an online, English survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult self-identified minorities (African, Asian, Hispanic/Latino, American Indian, Alaskan native, etc.)
Sampling Method: Probability Sample
Enrollment: 619 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Frequency of skin tone differences between ideal and actual | 6 months
  The frequency at which research participants indicate ideal skin tone differences versus actual will be assessed in the questionnaire. The unit of measure will be a numerical value, number of participants.

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University Feinberg School of Medicine Department of Dermatology, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No